CLINICAL TRIAL: NCT00005951
Title: Phase I Treatment of Adults With Primary Malignant Glioma With Irinotecan (CPT-11) (NSC- #6616348) Plus Temodar (NSC #362856)
Brief Title: Irinotecan Plus Temozolomide in Treating Patients With Recurrent Primary Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 1087; DUMC-1087-02-6R3; DUMC-001087-006R1; DUMC-1067-99-6; NCI-G00-1795; DUMC-001087-01-6R2; CDR0000067931
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Gliosarcoma | interventions — Irinotecan; Temozolomide

INTERVENTIONS:
Drug: irinotecan hydrochloride
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of irinotecan plus temozolomide in treating patients who have recurrent primary malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of irinotecan administered in combination with temozolomide in patients with recurrent primary malignant glioma.
* Determine the toxicity of this combination therapy in these patients.

OUTLINE: This is a dose escalation study of irinotecan. Patients are stratified according to concurrent anticonvulsants (Dilantin, Tegretol, or phenobarbital vs other anticonvulsants or none).

Patients receive irinotecan IV over 90 minutes on days 1, 8, 15, and 22 and oral temozolomide on days 1-5. Treatment continues every 43 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent primary malignant glioma

  * Anaplastic astrocytoma
  * Glioblastoma multiforme
  * Anaplastic oligodendroglioma
  * Gliosarcoma
  * Anaplastic mixed oligoastrocytoma
* Measurable disease by MRI or CT
* No immediate radiotherapy required
* Neurologically stable for at least 2 weeks prior to study

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Greater than 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT and SGPT less than 2.5 times ULN
* Alkaline phosphatase less than 2 times ULN

Renal:

* Blood urea nitrogen and creatinine less than 1.5 times ULN

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No other nonmalignant systemic disease
* No acute infection treated with IV antibiotics
* No frequent vomiting or other condition that would preclude oral medication administration (e.g., partial bowel obstruction)
* No other prior malignancies except surgically cured carcinoma in situ of the cervix or basal or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No more than 1 prior biologic therapy regimen

Chemotherapy:

* No more than 1 prior chemotherapy regimen
* At least 6 weeks since prior chemotherapy, unless evidence of disease progression
* No prior failure of irinotecan or temozolomide

Endocrine therapy:

* Concurrent corticosteroids allowed

Radiotherapy:

* See Disease Characteristics
* At least 6 weeks since prior radiotherapy, unless evidence of disease progression

Surgery:

* At least 3 weeks since prior surgery, unless evidence of disease progression, and recovered

Other:

* No concurrent immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States